CLINICAL TRIAL: NCT02729870
Title: Oral Glucose Intervention for Children With Gastroenteritis and Ketosis
Status: Withdrawn | Type: Observational
Why Stopped: lack of funding
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201600147
Record Dates: First submitted 2016-03-29; First posted 2016-04-06 (Estimated); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Gastrointestinal Infections; Ketosis
Keywords: Ketones; Gastroenteritis
MeSH Terms: conditions — Ketosis; Gastroenteritis | interventions — Carboxymethylcellulose Sodium; Gels

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Oral Glucose Gel: This group will consist of participants ages 1 - 7. The subject who are less than 3 year of age will receive 7.5 gram oral glucose gel 40% (0.66 oz, 20ml) which will be a one time dose and the subjects who are ages 3-7 will receive 15 gram oral glucose gel (1.3 oz, 40ml) which is a one time dose.
  Interventions: Drug: Oral Glucose Gel
- Oral Placebo Gel: The group will consist of participants ages 1 - 7. The subjects who are less than 3 years of age will receive carboxymethylcellulose (2%) oral gel, 20ml which will be a one time dose and the subjects ages 3- 7 will receive carboxymethylcellulose (2%) oral gel, 40ml which will be a one time dose.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Oral Glucose Gel — This group will receive the following: are less than 3 year of age will receive 7.5 gram oral glucose gel 40% (0.66 oz, 20ml) which will be a one time dose and the subjects who are ages 3-7 will receive 15 gram oral glucose gel (1.3 oz, 40ml) which is a one time dose.
  Other Names: Dextrose Gel; Glucote
  Groups: Oral Glucose Gel
Other: Placebo — This group will receive carboxymethylcellulose (2%) oral gel. The subjects who are less than than 3 years of age will receive carboxymethylcellulose (2%) oral gel, 20ml which will be a one time dose and the subjects ages 3-7 will receive carboxymethylcellulose (2%) oral gel, 40ml which will be a one time dose.
  Other Names: carboxymethylcellulose (2%) oral gel
  Groups: Oral Placebo Gel

SUMMARY:
Fasting ketoacidosis adds morbidity to children affected by gastrointestinal infections. The investigators investigate oral glucose gel for its effectiveness in rapidly reducing ketoacidosis and for improvements in oral hydration therapy success.

DETAILED DESCRIPTION:
More than 1.7 million children with acute gastroenteritis present for emergency department (ED) care annually in the United States. Gastroenteritis treatment regimens have been outlined in guidelines endorsed by the American Academy of Pediatrics, European Society of Pediatric Gastroenterology Hepatology and Nutrition (ESPGHAN), and Center for Disease Control (CDC). A fundamental principle included in these guidelines is the administration of oral rehydration therapy (ORT) to the vast majority of children with gastroenteritis; however, surveys have shown that a gap exists between guidelines and practice. Fasting ketoacidosis is an increasingly recognized metabolic derangement for children presenting with symptoms suggestive of gastroenteritis and mild to moderate dehydration. Ketoacidosis frequently occurs and likely adds comorbid symptoms of lethargy, vomiting, and malaise. These symptoms likely impair successful oral rehydration interventions. These symptoms may also lead to overestimations of the severity of dehydration. Rapid recognition of ketoacidosis is now possible with point of care testing beta-hydroxybutyrate. This investigation will determine if an oral glucose gel intervention will improve the Point Of Care (POC) beta-hydroxybutyrate from baseline. Secondary outcomes measured will include net fluid volume intake estimates, need for IV hydration, and need for hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Participants with gastroenteritis presenting to UF Health Shands Emergency Department

Exclusion Criteria:

* hypoglycemic- Blood glucose less than 50 or hyperglycemic- greater than 200

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged 1-7 years presenting to ED with symptoms of gastroenteritis
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-01 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Beta-hydroxybutyrate will be analyzed between the groups | Change from baseline to 4 hours
  Change in beta-hydroxybutyrate will be measured by blood test from -0 hour to 4 hours between the groups.

SECONDARY OUTCOMES:
The amount of oral fluid intake in milliliters will be measured between the groups | Change from 1 hour to 4 hours
  Oral fluid consumption will be measured between the groups.
Number of subjects Intravenous (IV)-Hydration between the groups | 4 hours
  Oral fluid hydration will have failed if subject needs IV fluid.
Number of subjects hospitalized between the groups | 4 hours
  The number of subjects with successful hydration can go home, however, the number of subjects who have to be hospitalized between the groups will be noted.

CONTACTS AND LOCATIONS:
Overall Officials: Fred R Guyer, MD, Principal Investigator — University of Florida Assisstant Professor

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Practice parameter: the management of acute gastroenteritis in young children. American Academy of Pediatrics, Provisional Committee on Quality Improvement, Subcommittee on Acute Gastroenteritis. Pediatrics. 1996 Mar;97(3):424-35. PMID 8604285
- [Background] Freedman SB, Steiner MJ, Chan KJ. Oral ondansetron administration in emergency departments to children with gastroenteritis: an economic analysis. PLoS Med. 2010 Oct 12;7(10):e1000350. doi: 10.1371/journal.pmed.1000350. PMID 20967234
- [Background] King CK, Glass R, Bresee JS, Duggan C; Centers for Disease Control and Prevention. Managing acute gastroenteritis among children: oral rehydration, maintenance, and nutritional therapy. MMWR Recomm Rep. 2003 Nov 21;52(RR-16):1-16. PMID 14627948
- [Background] Whyte LA, Al-Araji RA, McLoughlin LM. Guidelines for the management of acute gastroenteritis in children in Europe. Arch Dis Child Educ Pract Ed. 2015 Dec;100(6):308-12. doi: 10.1136/archdischild-2014-307253. Epub 2015 May 4. No abstract available. PMID 25939578
- [Background] Freedman SB, Gouin S, Bhatt M, Black KJ, Johnson D, Guimont C, Joubert G, Porter R, Doan Q, van Wylick R, Schuh S, Atenafu E, Eltorky M, Cho D, Plint A; Pediatric Emergency Research Canada. Prospective assessment of practice pattern variations in the treatment of pediatric gastroenteritis. Pediatrics. 2011 Feb;127(2):e287-95. doi: 10.1542/peds.2010-2214. Epub 2011 Jan 24. PMID 21262881
- [Background] Freedman SB, Thull-Freedman JD, Rumantir M, Atenafu EG, Stephens D. Emergency department revisits in children with gastroenteritis. J Pediatr Gastroenterol Nutr. 2013 Nov;57(5):612-8. doi: 10.1097/MPG.0b013e3182a1dd93. PMID 23820403
- [Background] Levy JA, Bachur RG, Monuteaux MC, Waltzman M. Intravenous dextrose for children with gastroenteritis and dehydration: a double-blind randomized controlled trial. Ann Emerg Med. 2013 Mar;61(3):281-8. doi: 10.1016/j.annemergmed.2012.08.007. Epub 2012 Sep 6. PMID 22959318
- [Background] Reid SR, Losek JD. Rehydration: role for early use of intravenous dextrose. Pediatr Emerg Care. 2009 Jan;25(1):49-52; quiz 53-4. doi: 10.1097/PEC.0b013e318191d97c. PMID 19148016
- [Background] Levy JA, Waltzman M, Monuteaux MC, Bachur RG. Value of point-of-care ketones in assessing dehydration and acidosis in children with gastroenteritis. Acad Emerg Med. 2013 Nov;20(11):1146-50. doi: 10.1111/acem.12256. PMID 24238317
- [Background] Harris DL, Weston PJ, Signal M, Chase JG, Harding JE. Dextrose gel for neonatal hypoglycaemia (the Sugar Babies Study): a randomised, double-blind, placebo-controlled trial. Lancet. 2013 Dec 21;382(9910):2077-83. doi: 10.1016/S0140-6736(13)61645-1. Epub 2013 Sep 25. PMID 24075361
- [Background] Barennes H, Valea I, Nagot N, Van de Perre P, Pussard E. Sublingual sugar administration as an alternative to intravenous dextrose administration to correct hypoglycemia among children in the tropics. Pediatrics. 2005 Nov;116(5):e648-53. doi: 10.1542/peds.2004-2218. PMID 16263979